CLINICAL TRIAL: NCT00021723
Title: Randomized Safety, Tolerability and Pilot Efficacy of AN-1792 in Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: JANSSEN Alzheimer Immunotherapy Research & Development, LLC (Industry)
Collaborators: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: VP Clinical Development, JANSSEN Alzheimer Immunotherapy Research & Development, LLC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AN-1792-201
Record Dates: First submitted 2001-08-02; First posted 2001-08-06 (Estimated); Last update posted 2009-09-24 (Estimated); Status verified 2001-11

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's; AN-1792; AIP-001
MeSH Terms: conditions — Alzheimer Disease

INTERVENTIONS:
Biological: AN-1792 also known as AIP-001

SUMMARY:
A multi-center, double-blind, placebo-controlled out-patient, safety, tolerability, and pilot efficacy study of intramuscular AN-1792 in patients with mild to moderate Alzheimer's disease.

DETAILED DESCRIPTION:
The study will enroll approximately 375 patients with mild to moderate Alzheimer's disease at investigational sites in the United States and Europe. Patients will receive either AN-1792 or placebo, and they will be evaluated using standard clinical assessments of cognition and memory as well as experimental surrogate markers of Alzheimer's disease pathology. The goal of the study is to evaluate the clinical impact of eliciting an immune response (formation of antibodies) to the A-beta peptide in patients with Alzheimer's disease.

ELIGIBILITY:
Mild to moderate Alzheimer's disease. Ability to cooperate with MRI scanning and neuropsychological testing. Live at home or in the community and a caregiver capable of accompanying the patient on all clinic visits and visiting the patient at least 5 times per week.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375
Dates: Start 2001-09; Study Completion 2003-09

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Pivotal Research Centers, Peoria, Arizona
  - 21st Century Neurology, Phoenix, Arizona
  - California Clinical Trials, Beverly Hills, California
  - UCSD Medical Center, La Jolla, California
  - Pharmacology Research Institute, Northridge, California
  - Baumel-Eisner Neuromedical Institute, Bay Harbor Islands, Florida
  - Baumel-Eisner Neuromedical Institute, Boca Raton, Florida
  - Baumel-Eisner Neuromedical Institute, Fort Lauderdale, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Clinical Pharmaceutical Trials, Inc., Tulsa, Oklahoma
  - Baylor College of Medicine, Houston, Texas